CLINICAL TRIAL: NCT02797106
Title: Management of Drooling in Children With Cerebral Palsy: A French Survey of the Practices and Opinions of Health Professionals
Brief Title: Management of Drooling in Children With Cerebral Palsy in France
Acronym: TOXSIALO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D21660
Record Dates: First submitted 2016-05-31; First posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: Cerebral Palsy; Pathological Drooling
Keywords: Drooling; Cerebral palsy; Botulinium toxin; Practice survey of health professionals; Children
MeSH Terms: conditions — Cerebral Palsy; Sialorrhea

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- health care professionals: health care professionals potentially involved in assessment and/or treatment of drooling in children with Cerebral Palsy.
  Interventions: Other: Practice survey of health professionals

INTERVENTIONS:
Other: Practice survey of health professionals — Survey of the practices and opinions of health care professionals to describe care pathways, assessment and treatment of drooling in children with cerebral palsy

SUMMARY:
The study is a transversal, observational, descriptive survey of the practices and opinions of health professionals carried out nationally across France that aims to characterize children with cerebral palsy and pathological drooling and to describe care pathways, assessment and treatment of drooling.

ELIGIBILITY:
Inclusion Criteria:

* health professional known to assess and/or treat drooling
* health professional known to assess and/or treat children with Cerebral Palsy
* health professional exercising in France

Exclusion Criteria:

* health professional with an inactive e-mail address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: health care professionals potentially involved in assessment and/or treatment of drooling in children with Cerebral Palsy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Questionnaire on the assessment and treatment of drooling in children with Cerebral Palsy | Day 1 (At the time of the questionnaire mailing to the professionals)
  Questionnaire will measure practices of health professionals involved in care pathways, assessment and treatment of drooling in children with Cerebral Palsy.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle CHALEAT-VALAYER, MD, Principal Investigator — CMCR des Massues -Croix Rouge Française, Lyon